CLINICAL TRIAL: NCT01674946
Title: Effect of Intraduodenal Perfusion of Bile Acids on the Secretion of Gastrointestinal Satiation Peptides in Healthy Male Volunteers
Brief Title: Effect of Bile Acids on the Secretion of Satiation Peptides in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 140/11
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Echolocation
Keywords: GI-physiology; CDCA; bile acids; TGR5; satiation peptides
MeSH Terms: conditions — Echolocation | interventions — Sodium Chloride; Bile Acids and Salts; Chenodeoxycholic Acid; Oleanolic Acid; Oleic Acid; Fatty Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ID saline (Placebo Comparator): ID saline by feeding tube
  Interventions: Other: saline
- ID saline + CDCA (5 mmol/L) (Active Comparator): CDCA = chenodeoxycholic acid (primary bile acid)
  Interventions: Other: saline; Other: bile acid (CDCA, chenodeoxycholic acid)
- ID + CDCA (15 mmol/L) (Active Comparator): CDCA = chenodeoxycholic acid (primary bile acid)
  Interventions: Other: saline; Other: bile acid (CDCA, chenodeoxycholic acid)
- ID saline + oleanolic acid (1 mmol/L) (Active Comparator)
  Interventions: Other: saline; Other: oleanolic acid
- ID saline + CDCA (5 mmol/L) + oleic acid (Active Comparator)
  Interventions: Other: saline; Other: bile acid (CDCA, chenodeoxycholic acid); Dietary Supplement: oleic acid
- ID saline + oleic acid (20 mmol/L) (Placebo Comparator)
  Interventions: Other: saline; Dietary Supplement: oleic acid

INTERVENTIONS:
Other: saline — intraduodenal perfusion
Other: bile acid (CDCA, chenodeoxycholic acid) — intraduodenal perfusion
  Other Names: primary bile acid
  Arms: ID + CDCA (15 mmol/L); ID saline + CDCA (5 mmol/L); ID saline + CDCA (5 mmol/L) + oleic acid
Other: oleanolic acid — intraduodenal perfusion
  Other Names: triterpenoid compound of plant origin
  Arms: ID saline + oleanolic acid (1 mmol/L)
Dietary Supplement: oleic acid — intraduodenal perfusion
  Other Names: fatty acid
  Arms: ID saline + CDCA (5 mmol/L) + oleic acid; ID saline + oleic acid (20 mmol/L)

SUMMARY:
The purpose of this study is do determine the functional significance of the G protein-coupled receptor TGR5 in the secretion of GI satiation peptides by using natural bile acids and oleanolic acid (triterpenoid compound of plant origin) as TGR5 agonists.

DETAILED DESCRIPTION:
TGR5 is expressed in GLP-1-secreting cell lines and L cells from mice; gain- and loss-of-function models suggest a physiological role for TGR5 activation on GLP-1 secretion in rodents. TGR5 signaling showed improved postprandial glucose tolerance in obese mice, associated with marked postprandial GLP-1 release and insulin secretion. In contrast, TGR5-/- mice exhibited reduced glucose tolerance. In animals, TGR5 activation has been shown for natural bile acids (BAs) and triterpenoid compounds of plant origin, such as oleanolic acid (OA), suggesting a role for postprandial BAs in modulating nutrient-induced GLP-1 secretion. We therefore hypothesized that intraduodenal (ID) perfusions of TGR5 agonists (BAs and OA) stimulate the secretion of GLP-1 with respective changes in the glucose metabolism of healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* BMI of 19.0-24.5
* Age 18-40
* Stable body weight for at least 3 months

Exclusion Criteria:

* Smoking
* Substance abuse
* Regular intake of medication
* Medical of psychiatric illness
* Gastrointestinal disorders or food allergies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal satiation peptide secretion | 3 hours blood sampling
  Assessment of plasma GLP-1, PYY and CCK release to BA and OA stimulation

SECONDARY OUTCOMES:
Serum bile acids | 3 hours blood sampling
  Assessment of serum bile acids levels to BA and OA stimulation
Appetite perceptions during 3 hours using visual analogue scales | 3 hours
  Assessment of the following appetite perceptions markers: feelings of hunger, feelings of prospective food consumption, feelings of fullness and feelings of satiety using validated visual analogue scales
Glucose and insulin secretion | 3 hours blood sampling
  Assessment of plasma glucose and insulin levels to BA and OA stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital Basel, Phase 1 Research Unit, Basel Switzerland
Locations (1):
- University Hospital Basel, Phase 1 Research Unit, Basel, Switzerland